CLINICAL TRIAL: NCT03537443
Title: Effect of Maternal Vitamin D Supplementation During Pregnancy on Offspring Bone Mass, Body Composition and Muscle Strength in Early Childhood: Follow-up of a Randomized Controlled Trial Cohort.
Brief Title: Bone and Muscle Health in Kids
Acronym: BONUSKids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Daniel Roth, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1000060961
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Skeletal Disorder
Keywords: Childhood; Vitamin D; Bone mineral density; Bone mineral content
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A (Placebo) (Placebo Comparator): Children whose mothers were randomized to receive a weekly dose of placebo from 17-24 weeks of gestation to 26 weeks postpartum.
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3)
- Group B (4200:0 IU/week) (Experimental): Children whose mothers were randomized to receive a prenatal:postpartum regimen of 4200 IU/week vitamin D3 from 17-24 weeks of gestation to delivery, followed by placebo from delivery to 26 weeks postpartum.
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3)
- Group C (16800:0 IU/week) (Experimental): Children whose mothers were randomized to receive a prenatal:postpartum regimen of 16800 IU/week vitamin D3 from 17-24 weeks of gestation to delivery, followed by placebo from delivery to 26 weeks postpartum.
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3)
- Group D (28000:0 IU/week) (Experimental): Children whose mothers were randomized to receive a prenatal:postpartum regimen of 28000 IU/week vitamin D3 from 17-24 weeks of gestation to delivery, followed by placebo from delivery to 26 weeks postpartum.
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3)
- Group E (28000:28000 IU/week) (Experimental): Children whose mothers were randomized to receive a prenatal:postpartum regimen of 28000 IU/week vitamin D3 from 17-24 weeks of gestation to delivery, followed by the same dose (28000 IU/week vitamin D3) from delivery to 26 weeks postpartum.
  Interventions: Dietary Supplement: Cholecalciferol (vitamin D3)

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (vitamin D3) — Prenatal and postpartum supplementation with vitamin D3 and/or placebo.

SUMMARY:
Vitamin D deficiency in childhood leads to poor bone growth and muscle weakness, yet it is unknown if the amount of vitamin D a woman consumes during her pregnancy affects her child's bone and muscle development. In collaboration with researchers in Bangladesh, the investigators recently completed a study of vitamin D supplementation during pregnancy in which women were assigned to 1 of 5 groups containing vitamin D or placebo (no vitamin D). The investigators now aim to conduct a follow-up study of a sample of 600 4 year old children born to these mothers to test the possible effects of vitamin D supplementation in pregnancy on children's bones, their body composition and the strength of their muscles.

DETAILED DESCRIPTION:
Vitamin D is a modifiable regulator of bone mineral metabolism and muscle function; yet little is known about the role of in utero vitamin D exposure on bone mineral accrual and muscle development in early childhood. Observational findings suggest associations between prenatal vitamin D status and infant bone, lean and fat mass and muscle function, but data from intervention trials is either unavailable or limited to early infancy. The investigators of the proposed study have previously shown that prenatal vitamin D supplementation safely improves maternal-fetal vitamin D status and perinatal calcium metabolism. Given the current interest in the potential role of vitamin D in perinatal health, adequately powered and well-designed randomized trials are required to investigate the effect of maternal vitamin D supplementation on offspring musculoskeletal health and body composition.

The investigators recently conducted the Maternal Vitamin D for Infant Growth (MDIG) trial (NCT01924013), a randomized placebo-controlled dose-ranging trial of vitamin D supplementation in pregnancy and lactation in Bangladesh, where severe vitamin D deficiency is common. Women at 17-24 weeks' gestation were randomized to 1 of 5 dose groups comprising a prenatal:postpartum regimen of placebo:placebo, 4200:0, 16800:0, 28000:0 or 28000:28000 IU vitamin D3/week until 26 weeks postpartum. Enrolment (n=1300) was completed in September 2015, and all infants were delivered by February 2016. The MDIG trial was primarily designed to determine the effect of maternal vitamin D on infant length at 12 months of age, with follow-up continuing until infants reached 24 months of age (completed in March 2018).

In the proposed observational follow-up study, the investigators will leverage the design and infrastructure of the MDIG trial to investigate effects of vitamin D on early childhood bone and muscle outcomes in a sample of MDIG participants at 4 years of age (target n=600 with 120 participants per maternal vitamin D treatment group; to allow for an expected attrition rate of 15%, the required sample size will be inflated to 140 children per group, giving an overall target sample size of 700 children).

The primary objective is to quantify the effects of prenatal vitamin D supplementation versus placebo on offspring total-body-less head (TBLH) bone mineral content and density. Secondary objectives are to examine the effect of vitamin D on TBLH lean and fat mass, and muscle function. Bone, lean and fat mass will be measured using dual-energy x-ray absorptiometry (DXA). Muscle strength (handgrip test), anthropometry, dietary intake and vitamin D status will also be assessed, in addition to biomarkers of bone turnover that may affect musculoskeletal health in young children.

The proposed follow-up study of a large randomized trial will contribute new evidence regarding the effects of vitamin D supplementation during pregnancy on musculoskeletal health in childhood.

Data analysis

Owing to the large contribution of head BMC values to whole-body BMC, in addition to difficulties in obtaining accurate head positioning without motion artifact in young children, TBLH BMC will be considered as the primary outcome in the present study. While TBLH BMC and TBLH areal BMD are closely related and complementary measures of bone mass, and both will be examined in the main analyses, TBLH BMC will be considered as the primary outcome measure. Whole-body measurements will be examined as secondary outcomes, in addition to BMC and areal BMD measurements of the head alone. DXA-derived estimates of lean and fat mass will also first be explored as TBLH measures, and later explored as whole-body measurements. Primary analyses will be conducted without adjustment for covariates; however, adjustment for concurrent body size, age or child sex will be explored in additional analyses.

Placebo versus high-dose prenatal vitamin D supplementation: To address the objectives with maximum statistical efficiency, the 2 high-dose prenatal vitamin D groups will be combined for a comparison of children of mothers who received 28000 IU/week of vitamin D prenatally (with or without 28000 IU/week of vitamin D postpartum) versus those children whose mothers received placebo prenatally. Differences will be expressed as mean differences with 95% CIs, and tested for statistical significance using t-tests. In sub-group analyses, we will stratify by baseline maternal vitamin D status (25(OH)D ≥ 30 nmol/L vs < 30 nmol/L) or infant sex (boys vs girls). A restricted analysis will also be completed, limited to term-born infants only (≥37 weeks' gestation).

Dose-response effect of prenatal and postpartum vitamin D supplementation: For the dose-response analysis including data from all treatment groups, we will regress each outcome (as a continuous variable) on the assigned dose of vitamin D (as a categorical variable) during the prenatal period (with the 2 high-dose prenatal vitamin D treatment groups combined). In this way, mean differences of each prenatal supplementation group will be compared to the placebo group, to test the effect of prental supplementation only. We will also regress each outcome on the average weekly dose of vitamin D assigned as a continuous variable during the prenatal period. Similar regression models will be conducted using more precise estimates of the vitamin D dose received, based on manufacturer analysis of the vitamin D composition of each batch of tablets provided and individual compliance with study tablets. We will use linear regression splines to accommodate non-linear outcome-dose relationships if warranted based on non-parametric visualization (e.g. LOWESS). To ensure precision of the 95% CIs, and therefore ensure robust inferences, 95% CIs from the linear regression models will be obtained using bootstrapping (with 1000 replications).

To explore potential effects of prenatal only versus prenatal plus postpartum vitamin D supplementation, a similar dose-response analysis will be conducted across all 5 treatment groups (i.e., disaggregation of the 2 high-dose prenatal vitamin D groups), for which we will regress each outcome (as a continuous variable) on the vitamin D treatment group assigned during the prenatal and postpartum periods (as a categorical variable). Mean differences of each supplementation group will therefore be compared to the placebo group. Estimates of the 95% CIs from all regression models will be obtained using bootstrapping (with 1000 replications).

Further exploratory analyses of primary and secondary outcomes: Multivariable regression models will enable adjustment for other potential determinants of bone mass, muscle function and body composition including: baseline covariates that differed by treatment group (if present) and thus may confound treatment effects; child characteristics at the time of assessment (e.g. vitamin D status); maternal characteristics (e.g. education level) and socioeconomic status of the household. We will include measures of height or weight (e.g., height-for-age Z-scores) as covariates to test their roles in mediating the effect of the vitamin D intervention on bone mass or other outcomes (muscle strength, body composition). Linear regression models will also be used to assess between-group differences in calcium metabolism and bone turnover markers.

ELIGIBILITY:
Inclusion Criteria:

The sample population will be drawn from a cohort registry of mother-infant pairs who participated in the recently-completed Maternal Vitamin D for Infant Growth (MDIG) randomized controlled trial (NCT01924013):

* Child is available for participation at 45 to 51 months postnatal age
* Mother received ≥80% of assigned prenatal vitamin D or placebo doses during the MDIG trial
* Child and primary caregiver(s) reside in Dhaka, Bangladesh or nearby regions
* A parent/guardian provides written or thumb-print informed consent for study procedures

Exclusion Criteria:

* Mother participated in the MDIG trial but chose not to be included in the cohort registry for contact regarding follow-up studies
* Children outside the eligible age range (aged below 45 months or above 51 months)
* Child is diagnosed with any developmental disorder that would render difficulty in completion of the DXA scan (e.g. Autism)
* Child is unable to bear weight on his/her legs (e.g. wheelchair bound)
* Child has a current fracture or break in which his/her limb is supported by an orthopedic cast

Ages: 45 Months to 51 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 642 (Actual)
Dates: Start 2018-10-21 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Total-body-less head bone mineral content and total-body-less head bone mineral density | 4 years of age
  Measured by DXA

SECONDARY OUTCOMES:
Muscle function (handgrip strength) | 4 years of age
  Measured by hand-held dynamometer
Total-body-less head lean and total-body-less head fat mass | 4 years of age
  Measured by DXA
Whole-body (including head) bone mineral content and whole-body bone mineral density | 4 years of age
  Measured by DXA
Head bone mineral content and head bone mineral density | 4 years of age
  Measured by DXA
Whole-body lean and whole-body fat mass | 4 years of age
  Measured by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- International Center for Diarrheal Disease Research, Dhaka, Bangladesh

REFERENCES:
- [Derived] O'Callaghan KM, Funk C, Fariha F, Nagaria MH, Dasiewicz A, Harrington J, Mahmud AA, Abrams SA, Ahmed T, Moore DR, Roth DE. Serum 25-Hydroxyvitamin D and Intact Parathyroid Hormone as Functional Biomarkers of Bone Mass in Early Childhood. J Nutr. 2025 Jun;155(6):1782-1794. doi: 10.1016/j.tjnut.2025.03.022. Epub 2025 Mar 24. PMID 40139482
- [Derived] O'Callaghan KM, Shanta SS, Fariha F, Harrington J, Mahmud AA, Emdin AL, Gernand AD, Ahmed T, Abrams SA, Moore DR, Roth DE. Effect of maternal prenatal and postpartum vitamin D supplementation on offspring bone mass and muscle strength in early childhood: follow-up of a randomized controlled trial. Am J Clin Nutr. 2022 Mar 4;115(3):770-780. doi: 10.1093/ajcn/nqab396. PMID 34849536